CLINICAL TRIAL: NCT00776867
Title: Phase I Study of Single Agent Perifosine for Recurrent Pediatric Solid Tumors
Brief Title: Study of Single Agent Perifosine for Recurrent Pediatric Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Wisconsin, Madison (Other); Duke University (Other); AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-091
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumors
Keywords: Pediatric; solid tumors; Pediatric solid tumors; 08-091
MeSH Terms: interventions — perifosine

ARMS (1):
- perifosine (Experimental): This will be a dose escalation study to determine the maximum tolerated dose (MTD) of perifosine alone in recurrent/progressive pediatric tumors. A standard 3+3 dose escalation design will be employed with 3-6 patients at each dose level.
  Interventions: Drug: perifosine

INTERVENTIONS:
Drug: perifosine — Open label, phase I study of oral perifosine in recurrent/progressive pediatric solid tumors. This will be a dose escalation study to determine the maximum tolerated dose (MTD) of perifosine alone in recurrent/progressive pediatric tumors. A standard 3+3 dose escalation design will be employed with 3-6 patients at each dose level. All patients will receive perifosine at a loading dose on the first day, followed by a maintenance dose to start on day two until progression each patient will be assigned to a dosing group based on one's body surface area (BSA).

SUMMARY:
The purpose of this study is to test whether perifosine- a drug that inhibits the protein AKT, and has had some success in the treatment of adult cancers- is safe and effective in treating cancer. The investigators want to find out what effects, good and/or bad, it has on the patient and the cancer. The investigators are testing different dose schedules of perifosine and the patient will be asked to partake in one of the dose schedules.

ELIGIBILITY:
Inclusion Criteria:

* Any solid tumor that failed standard therapy.
* Patient must have evidence for tumor by CT, MRI, PET scan, MIBG scan, serum markers, or tissue sampling.
* Age ≤ 21 years.
* Karnofsky/Lansky performance status ≥ 50% (Karnofsky score for age> 16 years and Lansky score for age ≤ 16 years)
* ANC≥ 1000 at least 24 hours off GCSF
* Platelets ≥ 75k at least one week off platelet transfusions
* Hg≥ 8g/dL at least one week off PRBC transfusion
* AST ≤ 3 x the upper limit of normal
* ALT ≤ 3 x the upper limit of normal
* Total bilirubin ≤ 2.0 mg/dl
* serum creatinine ≤ 1.5 x the upper limit of normal for age, or calculated creatinine clearance or nuclear GFR ≥ 70 ml/min/1.73 m2.
* ≥ 3 weeks since last non-nitrosourea chemotherapy
* ≥ 6 weeks since last nitrosoureas
* ≥ 4 weeks since last RT
* Patients must agree to practice adequate contraception. Females of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to drug initiation. Females must not be breast feeding.
* Patients must be able to swallow tablets whole

Exclusion Criteria:

* Pregnancy
* Patients must not have active infection or serious intercurrent medical illness.
* HIV-Positive patients receiving combination anti-retroviral therapy are excluded from the study due to possible retro-viral drug interactions. HIV testing not required.
* Patients must not be taking EIAEDs. If patients were previously EIAEDs that have been discontinued, patients must have been off the agent for at least 2 weeks prior to registration.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2008-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of perifosine monotherapy in children with cancer | conclusion of the study

SECONDARY OUTCOMES:
To determine whether pharmacokinetic serum levels correlate with toxicity | conclusion of the study
If previously resected tissue is available, determine whether molecular features predict response including Elevated PI3K/AKT/mTOR signaling, Elevated RAS/MAPK signaling, Cell cycle markers | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Cheung NV, Modak S, Becher OJ, Basu EM, Roberts SS, Kramer K, Dunkel IJ. A phase I/Ib trial targeting the Pi3k/Akt pathway using perifosine: Long-term progression-free survival of patients with resistant neuroblastoma. Int J Cancer. 2017 Jan 15;140(2):480-484. doi: 10.1002/ijc.30440. Epub 2016 Sep 30. PMID 27649927
- [Derived] Sun W, Modak S. Emerging treatment options for the treatment of neuroblastoma: potential role of perifosine. Onco Targets Ther. 2012;5:21-9. doi: 10.2147/OTT.S14578. Epub 2012 Mar 2. PMID 22419878
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org